CLINICAL TRIAL: NCT02571088
Title: Evaluation of a Training Program for Homozygous Sickle Cell Disease Patients: Benefits on Physical Ability and Skeletal Muscle. An Interventional Pilot, Multicentric, Prospective, Longitudinal Study
Brief Title: Evaluation of a Training Program for Homozygous Sickle Cell Disease Patients
Acronym: EXDRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Centre de Référence des Syndromes Drépanocytaires Majeurs (Other); Laboratoire de Physiologie de l'Exercice (Unknown); Claude Bernard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1408030; 2014-A00334-43 (Other: ANSM)
Record Dates: First submitted 2015-08-25; First posted 2015-10-08 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Sickle Cell Hemoglobin C Disease; Hemoglobin S Disease
Keywords: Sickle Cell Hemoglobin C Disease; Sports Training; Hemoglobin S Disease; Lactate
MeSH Terms: conditions — Hemoglobin SC Disease; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training Program (Experimental): The treatment will consist in an endurance training program. Only patients of the trained group will be subjected to this training program which will typically consist in 3 training sessions per week during 8 weeks i.e., 24 training sessions. Each training session will last 45 min. All training sessions will take place at the hospital and will be under medical supervision.
  Interventions: Other: Training Program
- No Training Program (No Intervention): It will be asked to the control patients to not change their habitual physical activity during the entire period of observation

INTERVENTIONS:
Other: Training Program — Each training session will last 45 min. Exercise will start by a 5-min warm-up cycling period, followed by 30 min of cycling at the power output (W) individually determined before and corresponding to the first lactate threshold corresponding approximately to 2.5 mmol/l . Then patients will cool down for 5 min. Finally, the training sessions will end by 5 min of light stretching. All training sessions will take place at the hospital and will be under the supervision of a physician. Heart rate, oxygen saturation and blood lactate concentrations will be regularly measured. Work rate will be adjusted according to the obtained results. As a safety procedure, blood lactate concentration must not exceed 4 mmol/L during the training sessions. A particular attention will be paid to the hydration of patients. Pain and fatigue will be evaluated everyday by the patients using (100 mm) visual analog scales.
  Arms: Training Program

SUMMARY:
Sickle cell disease (SCD) is the most frequent inherited disease in the world. Literature reports that SCD patients display intolerance to exercise, important muscle weakness and profound remodeling of skeletal muscle including amyotrophy and rarefied microvascular network.

Because strenuous exercise induces acidosis, hemorheological alterations, endothelial activation and oxidative stress, it constitutes a potential triggering factor of sickling and vaso-occlusive crisis. As a consequence, physical activity is usually discouraged in patients with SCD. However, moderate and regular physical activity seems to be not only safe but also beneficial for SCD patients.

DETAILED DESCRIPTION:
Besides, endurance training is known to induce moderate muscle hypertrophy and increase microvascular network. Therefore, adapted, moderate and regular physical activity appears as a potential strategy able to improve muscle function, decrease symptoms of the disease and improve autonomy and quality of life of patients with SCD. However, it remains necessary to define the modalities of exercise therapy in SCD and to objectively evaluate the risks, limitations and gains on physical ability, muscle function and quality of life in patients with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease patient (HbSS or HbS-βthal0),
* Affiliated to a Health Security program,
* Consent form signed,
* Patients in stabilized state at the onset of the experiment: at least one month after an acute adverse event and at least 3 months after a blood transfusion.

Exclusion Criteria:

* Patients whom adhesion/compliance to the protocol appears uncertain,
* Patient involved in another clinical trial or within the exclusion period of a previous clinical trial,
* Patients known to be affected by a chronic inflammatory or infectious pathology,
* Patients having an intercurrent infection, especially inflammatory, unsolved since less than one month,
* Patients with clinical signs of heart failure or hospitalized for cardiac decompensation during the past 12 months,
* Patients with left ventricular ejection fraction < 50%, pulmonary arterial hypertension with tricuspid regurgitation velocity > 2.5 m/s, atrial fibrillation, ventricular rhythm disorders during exercise, left ventricular hypertrophy (septal to lateral wall thickness ≥ 10 mm), significant valvulopathy, established coronary disease, uncontrolled hypertension,
* Patients with a treatment against cardiac arrhythmia or altering sino-atrial node activity (beta-blockers, atropine, sympathomimetic agents…),
* Patients under anti-coagulant treatment,
* Patients with pacemaker or defibrillator,
* Body Mass Index (BMI) > 35,
* Patients with hip osteonecrosis,
* Patients with cerebral vasculopathy or history of stroke (cerebrovascular attack) with epilepsy,
* Pregnant or lactating patients,
* Homeless patients,
* Patients with the inability to understand the aims,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Power output (W) associated with the 4 mmol/L blood lactate concentration | 8 weeks
  The blood lactate concentration curve in response to incremental exercise depends on the physical ability of patients. Endurance training is known to increase the power output (W) associated with a given blood lactate concentration. For the present study, we used the 4 mmol/L blood lactate concentration as a remarkable/singular point of the curve

SECONDARY OUTCOMES:
Muscle fiber types distribution (%) | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
perimeter (µm) of muscle fiber | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
surface area (µm2) of muscle fiber | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
satellite cell account | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
Creatine Kinase (CK) of muscle | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
Phosphofructokinase (PFK) of muscle | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
Citrate Synthetase (CS) of muscle | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
HAD (µmol/min/g dry muscle) of muscle | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
COx (arbitrary unit, a.u.) of muscle | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
Lactate Dehydrogenase (LDH) of muscle | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
isoforms (%) of muscle | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
Number of capillaries per mm2 (capillary density) and in contact with a muscle fiber | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
surface area of microvessels (µm2) | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
diameter of microvessels (µm) | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
capillary tortuosity (quotient) | 8 weeks
  Patients will be subjected to a biopsy of the vastus lateralis muscle (≈ 200 mg).
expired volume (VE) | 8 weeks
  Patients will perform a submaximal incremental exercise on a cycle ergometer. Exercise will start at 20 W and 30 W for females and males, respectively. After 2 minutes at this load, and every 2 minutes thereafter, work rate will increase by 10 W and 15 W for females and males, respectively. Total exercise duration is expected to be within 8 to 14 minutes.
oxygen consumption (VO2) | 8 weeks
  Patients will perform a submaximal incremental exercise on a cycle ergometer. Exercise will start at 20 W and 30 W for females and males, respectively. After 2 minutes at this load, and every 2 minutes thereafter, work rate will increase by 10 W and 15 W for females and males, respectively. Total exercise duration is expected to be within 8 to 14 minutes.
carbon dioxide production (VCO2) (L/min) | 8 weeks
  Patients will perform a submaximal incremental exercise on a cycle ergometer. Exercise will start at 20 W and 30 W for females and males, respectively. After 2 minutes at this load, and every 2 minutes thereafter, work rate will increase by 10 W and 15 W for females and males, respectively. Total exercise duration is expected to be within 8 to 14 minutes.
respiratory quotient (QR) | 8 weeks
  Patients will perform a submaximal incremental exercise on a cycle ergometer. Exercise will start at 20 W and 30 W for females and males, respectively. After 2 minutes at this load, and every 2 minutes thereafter, work rate will increase by 10 W and 15 W for females and males, respectively. Total exercise duration is expected to be within 8 to 14 minutes.
Heart Rate (HR) (min-1) | 8 weeks
  Patients will perform a submaximal incremental exercise on a cycle ergometer. Exercise will start at 20 W and 30 W for females and males, respectively. After 2 minutes at this load, and every 2 minutes thereafter, work rate will increase by 10 W and 15 W for females and males, respectively. Total exercise duration is expected to be within 8 to 14 minutes.
lactate level (mmol/l) at the end of submaximal incremental exercise | 8 weeks
  Patients will perform a submaximal incremental exercise on a cycle ergometer. Exercise will start at 20 W and 30 W for females and males, respectively. After 2 minutes at this load, and every 2 minutes thereafter, work rate will increase by 10 W and 15 W for females and males, respectively. Total exercise duration is expected to be within 8 to 14 minutes.
Pulmonary volumes (L) | 8 weeks
  The volumes are measured by plethysmography
Performance to the six minute walk test (m) | 8 weeks
Index of muscular blood flow and tissular oxygenation at rest (%) | 8 weeks
  Patients will perform a submaximal incremental exercise on a cycle ergometer. Exercise will start at 20 W and 30 W for females and males, respectively. After 2 minutes at this load, and every 2 minutes thereafter, work rate will increase by 10 W and 15 W for females and males, respectively. Total exercise duration is expected to be within 8 to 14 minutes.
Index of exercise using Near-infrared reflectance spectroscopy (NIRS) (%) | 8 weeks
  Patients will perform a submaximal incremental exercise on a cycle ergometer. Exercise will start at 20 W and 30 W for females and males, respectively. After 2 minutes at this load, and every 2 minutes thereafter, work rate will increase by 10 W and 15 W for females and males, respectively. Total exercise duration is expected to be within 8 to 14 minutes.
Maximal voluntary contraction (N) | 8 weeks
  Maximal Voluntary Contraction (MVC) will be measured 3 times 1 min apart to determine an initial MVC. After 10 min of rest following the MVC trials, neuromuscular fatigability will be assess by repetition of series of 10 submaximal contractions (of 4 s separated by 5 s) followed by a MVC trial until a decrease of 25% of the initial MVC is observed. No more than 7 series will be performed, even if the 25% decrease of initial MVC is not observed.
Neuromuscular fatigability (%) | 8 weeks
  It is measured in the same time that MVC
Quality of life : Scores to the Short Form 36 (SF-36) | 8 weeks
Quality of life : Functional Assessment of Cancer Therapy (FACT Fatigue Part) | 8 weeks
Quality of life : State-Trait Anxiety Scale (STAI Y-A) | 8 weeks
Quality of life : Physical Self-Description Questionnaire( PSDQ) | 8 weeks
Complete blood count and biochemical analyses (ionogram, urea, creatinine, LDH, creatine phosphokinase (CPK), aspartate aminotransferase ; usual units) | 8 weeks
  Patients will be subjected to blood samplings
Blood and plasma viscosity (centipoise) | 8 weeks
  Patients will be subjected to blood samplings
Erythrocyte deformability (%) | 8 weeks
  Patients will be subjected to blood samplings
aggregation properties (a.u.) | 8 weeks
  Patients will be subjected to blood samplings
dense red blood cells (%) | 8 weeks
  Patients will be subjected to blood samplings
Plasma analyses of adhesion molecules and markers of inflammation | 8 weeks
  Patients will be subjected to blood samplings
oxidative stress | 8 weeks
  Patients will be subjected to blood samplings
NO metabolism (µmol/L) | 8 weeks
  Patients will be subjected to blood samplings
Activity of antioxidant enzymes (µmol/L/min) | 8 weeks
  Patients will be subjected to blood samplings
Expression of erythrocytes membrane proteins (u.a.) | 8 weeks
  Patients will be subjected to blood samplings
Red blood cell (RBC) adhesion to endothelial cells (count of adhering RBC /mm²) | 8 weeks
  Patients will be subjected to blood samplings
Various hemodynamic criteria using echocardiography at rest and exercise | 8 weeks
vaso-occlusive crises and acute chest syndrome | 8 weeks
  During the 8 weeks, all vaso-occlusive crises and acute chest syndrome will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Leonard FEASSON, MD, Principal Investigator — CHU de SAINT-ETIENNE; Laurent MESSONIER, PhD, Study Director — Université de Savoie
Locations (9):
- France (9):
  - Hopital Avicenne, Bobigny
  - Centre hospitalier sud francilien, Corbeil-Essonnes
  - CHU Henri MONDOR, Créteil
  - CHU Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - Hopital Europeen Georges POMPIDOU, Paris
  - Hopital Necker, Paris
  - Hopital Tenon, Paris
  - Centre hospitalier de Saint-Denis, Saint-Denis
  - CHU de SAINT-ETIENNE, Saint-Etienne

REFERENCES:
- [Derived] Merlet AN, Feasson L, Bartolucci P, Hourde C, Schwalm C, Gellen B, Galacteros F, Deldicque L, Francaux M, Messonnier LA; EXDRE Collaborative Study Group. Muscle structural, energetic and functional benefits of endurance exercise training in sickle cell disease. Am J Hematol. 2020 Nov;95(11):1257-1268. doi: 10.1002/ajh.25936. Epub 2020 Aug 1. PMID 32681734
- [Derived] Merlet AN, Messonnier LA, Coudy-Gandilhon C, Bechet D, Gellen B, Rupp T, Galacteros F, Bartolucci P, Feasson L. Beneficial effects of endurance exercise training on skeletal muscle microvasculature in sickle cell disease patients. Blood. 2019 Dec 19;134(25):2233-2241. doi: 10.1182/blood.2019001055. PMID 31742587
- [Derived] Gellen B, Messonnier LA, Galacteros F, Audureau E, Merlet AN, Rupp T, Peyrot S, Martin C, Feasson L, Bartolucci P; EXDRE collaborative study group. Moderate-intensity endurance-exercise training in patients with sickle-cell disease without severe chronic complications (EXDRE): an open-label randomised controlled trial. Lancet Haematol. 2018 Nov;5(11):e554-e562. doi: 10.1016/S2352-3026(18)30163-7. PMID 30389037